CLINICAL TRIAL: NCT05327855
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multiple-arm, Parallel-group, Adaptive Study to Investigate the Efficacy and Safety of OPL-0301 in Patients With Post-myocardial Infarction Left Ventricular Dysfunction (RESTORE)
Brief Title: Efficacy and Safety of OPL-0301 Compared to Placebo in Adults With Post-Myocardial Infarction (MI)
Acronym: RESTORE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn based on business decision, no participants enrolled
Sponsor: Valo Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPL-0301-201
Record Dates: First submitted 2021-12-22; First posted 2022-04-14 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Myocardial Infarction
Keywords: heart attack; acute ischemic heart disease; acute coronary syndrome; ST-Elevated Myocardial Infarction; left ventricular dysfunction
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Ventricular Dysfunction, Left

STUDY DESIGN:
Intervention Model Description: This is a Phase 2, multicenter, randomized, placebo-controlled, multiple-arm, adaptive study investigating the safety, pharmacokinetics, and potential efficacy of OPL-0301, along with standard of care, in post-myocardial infarction (MI) participants with left ventricular dysfunction (LVD).
  Participants will have been admitted to the hospital for acute MI and treated with primary percutaneous coronary intervention (PPCI) before entering the study. A fixed oral dose will be administered once daily, according to the blinded treatment assignment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OPL-0301 Dose 1 (Experimental): Participants are randomized to OPL-0301 Dose 1 administered once daily for 90 days
  Interventions: Drug: OPL-0301 Dose 1
- OPL-0301 Dose 2 (Experimental): Participants are randomized to OPL-0301 Dose 2 administered once daily for 90 days
  Interventions: Drug: OPL-0301 Dose 2
- Placebo (Placebo Comparator): Participants are randomized to matching placebo administered once daily for 90 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPL-0301 Dose 1 — Pharmaceutical form: Hard gelatin capsule; Route of administration: Oral
  Arms: OPL-0301 Dose 1
Drug: OPL-0301 Dose 2 — Pharmaceutical form: Hard gelatin capsule; Route of administration: Oral
  Arms: OPL-0301 Dose 2
Drug: Placebo — Pharmaceutical form: Hard gelatin capsule; Route of administration: Oral
  Arms: Placebo

SUMMARY:
Study OPL-0301-201 is intended to generate efficacy and safety data of OPL-0301 in participants with post-myocardial infarction (MI) left ventricular dysfunction (LVD)

DETAILED DESCRIPTION:
OPL-0301 is intended to address the disease state of post-myocardial infarction (MI) left ventricular dysfunction (LVD). MI is a manifestation of atherosclerotic coronary artery disease, the pathogenesis of which is closely associated with vascular and endothelial dysfunction, and inflammation. Acute MI leads to acute LVD, which often persists, leading to poor cardiovascular outcomes. The therapeutic hypothesis is that these effects mediated by Sphingosine-1 Phosphate 1 (S1P1) receptor agonism with OPL-0301 will reduce infarct size and benefit post-MI left ventricular function, thereby supporting improved cardiovascular outcomes in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female between 18 and 90 years of age, inclusive, at the time of signing the informed consent
* Are hospitalized with acute ST-Elevated Myocardial Infarction (STEMI), defined based on American Heart Association (AHA)/American College of Cardiology (ACC) criteria
* Have cardiac troponin-I (cTnI), cardiac troponin-T (cTnT) levels ≥10x upper limit of normal (ULN) at least once during the index event of myocardial infarction

Exclusion Criteria:

* Previous history of documented myocardial infarction
* Previous history of percutaneous coronary intervention (PCI) within 6 months or coronary artery bypass graft surgery (CABG) or valvular heart surgery at any time prior to screening
* Previous history of documented chronic left ventricular dysfunction with ejection fraction (EF) < 50%
* Previous history of decompensated heart failure
* Previous history of documented specific cardiomyopathy (including but not limited to hypertrophic cardiomyopathy (HCM), amyloid, sarcoid, etc.)
* Previous history of documented arrhythmias
* Are being treated with Sphingosine-1 Phosphate (S1P) modulators (fingolimod, siponimod, ozanimod, ponesimod)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Infarct size as determined by cardiac magnetic resonance (CMR) at Day 90 | 90 days
  To evaluate the effects of OPL-0301 versus placebo on infarct size in adults with post-myocardial infarction left ventricular dysfunction at day 90

SECONDARY OUTCOMES:
Change in infarct size by cardiac magnetic resonance (CMR) from initial CMR assessment to Day 90 | Initial to 90 days
  To evaluate the effects of OPL-0301 versus placebo on the change in infarct size in adults with post-myocardial infarction left ventricular dysfunction
Adverse events (AEs) and Serious adverse events (SAEs) | Baseline to 120 days
  To assess the effects of OPL-0301 on safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Victor Shi, M.D., Study Director — Valo Health, Inc.